CLINICAL TRIAL: NCT07173452
Title: The Effect of Women's Anthropometric Measurements on Pelvic Size and Labour Outcomes
Brief Title: Anthropometric Measurements on Size and Labour Outcomes
Acronym: Pelvis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Tuğba YILMAZ ESENCAN, Assistant Professor, Uskudar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023/06
Record Dates: First submitted 2025-07-01; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Pelvic Exam; Pelvis; Delivery Mode; Midwife
Keywords: Physical Body Measurements; External Pelvis Measurements; Labor Pain; Duration of Labor; Mode of Delivery; Midwife
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Intervention Model Description: This cross-sectional study was conducted between December 2022 and June 2023 in the labour ward of a maternity hospital in Istanbul and involved 153 pregnant women. The participants were evenly divided into three observational groups (arms), each consisting of 51 individuals, based on the method used to assess pelvic measurements. In the first group (Vaginal Examination Group), participants underwent pelvic assessment through standard vaginal examination techniques alongside physical body measurements. In the second group (External Pelvic Measurement Group), participants received external pelvic measurements using a pelvimeter in addition to physical body measurements. In the third group (Transvaginal Ultrasonographic Group), pelvic dimensions were evaluated via transvaginal ultrasonography along with physical body measurements. Each diagnostic approach served as the defining intervention for its respective group. Data were collected through face-to-face interviews and direct physical
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- the first group (Experimental): In the first group, participants' physical body measurements were evaluated alongside pelvic dimensions measured via vaginal examination.
  Interventions: Other: vaginal examination; Other: physical body measurements
- the second group (Experimental): In the second group, physical measurements were assessed together with external pelvic measurements.
  Interventions: Other: physical body measurements
- the third group (Experimental): In the third group, physical body measurements were evaluated in conjunction with pelvic assessments obtained through transvaginal ultrasonographic measurements.
  Interventions: Other: physical body measurements; Diagnostic Test: transvaginal ultrasonographic

INTERVENTIONS:
Other: vaginal examination — pelvic dimensions measured via vaginal examination.
  Arms: the first group
Other: physical body measurements — Anthrometric measurements of the participants were made
Diagnostic Test: transvaginal ultrasonographic — intrapartum pelvic evaluations were performed by transvaginal ultrasonography
  Arms: the third group

SUMMARY:
This study aims to evaluate women's physical body measurements and externally measurable pelvis measurements and determine their impact on labor pain level, duration of labor, and mode of delivery. The study was conducted between December 2022 and June 2023 at the Zeynep Kamil Women and Children's Health Education and Research Hospital in Istanbul, Turkey. The sample size was calculated using the OpenEpi program with a confidence interval of 80% and a sampling error of 0.05, resulting in a sample size of 139 individuals. Anticipating potential loss to follow-up during the study, the sample size was increased by 10% to 153 individuals. This sample group was divided into three equal groups, and pelvis measurement evaluations were recorded. Each group included 51 pregnant women. Data were collected through face-to-face measurements conducted by researchers using various forms, including an introductory information form, physical examination measurement form, transvaginal ultrasound measurement form, birth evaluation form, postpartum and neonatal evaluation form, visual analog pain scale (VAS) form, external pelvis measurement form and vaginal examination with pelvis measurement form.

DETAILED DESCRIPTION:
Background: One of the most critical factors in the progression of labour is the compatibility between the fetal head and the maternal pelvis. Therefore, the assessment of the pelvis during childbirth is of great importance.

Objectives: This study aims to evaluate women's physical body measurements in relation to externally measurable pelvic dimensions, to examine the relationship between them, and to determine their impact on pain levels during labour, the duration of labour, and the mode of delivery.

Methods: This cross-sectional study was conducted between December 2022 and June 2023 in the labour ward of a maternity hospital in Istanbul, involving 153 pregnant women. The sample was evenly divided into three groups, with 51 participants in each, and pelvic measurement assessments were recorded accordingly. In the first group, participants' physical body measurements were evaluated alongside pelvic dimensions measured via vaginal examination. In the second group, physical measurements were assessed together with external pelvic measurements. In the third group, physical body measurements were evaluated in conjunction with pelvic assessments obtained through transvaginal ultrasonographic measurements. The results obtained from the three groups were compared with one another. Data were collected through face-to-face interviews and direct measurements performed by the researchers using the following instruments: a descriptive information form, physical examination measurement form, transvaginal ultrasonography measurement form, labour assessment form, postpartum and neonatal evaluation form, visual analogue scale for pain, external pelvic measurement form, and vaginal pelvic examination form.

Keywords: Physical Body Measurements, External Pelvic Measurements, Labour Pain, Duration of Labour, Mode of Delivery, Midwife

ELIGIBILITY:
Inclusion Criteria:

* Primiparous,
* The onset of labour,
* Being between 37-42 weeks of gestation,
* To be able to speak and understand Turkish,
* 18 years of age or older,
* No history of a disease affecting bone anatomy

Exclusion Criteria:

* Risky pregnancies,
* Planned caesarean sections
* Multiparous pregnant women
* History of pelvic trauma, disease, previous pelvic surgeries.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women who gave birth constitute the sample of the study.
Enrollment: 153 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
vaginal examination | Measurements will be taken during the active phase of labor, when cervical dilation is between 4-10 cm (typically 6-12 hours prior to delivery), using a manual vaginal examination performed by an experienced obstetrician.
  Pelvic dimensions were evaluated by vaginal examination.
physical body measurements | Within the first 6 hours after the onset of active labor (defined as cervical dilation ≥4 cm).
  Maternal anthropometric parameters, including body weight (kg), height (cm), and Body Mass Index (BMI, kg/m²), will be assessed using standardized tools. Weight will be measured using a calibrated digital scale, and height using a calibrated stadiometer. BMI will be calculated using the formula:
  BMI = weight (kg) / [height (m)]².The weight and height will be combined to report BMI in kg/m^2.
transvaginal USG | Transvaginal ultrasonographic measurements will be performed within the first 2 hours after the onset of active labor, defined as cervical dilation ≥ 4 cm. These measurements will include fetal head position, angle of progression (in degrees), and head-p
  transvaginal ultrasonographic measurements

CONTACTS AND LOCATIONS:
Overall Officials: TUĞBA YILMAZ ESENCAN, Principal Investigator — TC Üsküdar Üniversitesi
Locations (1):
- Uskudar Univercity, Istanbul, Ümraniye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
starting in January 2026

REFERENCES:
- [Background] Benjamin SJ, Daniel AB, Kamath A, Ramkumar V. Anthropometric measurements as predictors of cephalopelvic disproportion: Can the diagnostic accuracy be improved? Acta Obstet Gynecol Scand. 2012 Jan;91(1):122-127. doi: 10.1111/j.1600-0412.2011.01267.x. Epub 2011 Oct 13. PMID 21895610
- See also: Anthropometric measurements as predictors of cephalopelvic disproportion: Can the diagnostic accuracy be improved? — https://pubmed.ncbi.nlm.nih.gov/21895610/